CLINICAL TRIAL: NCT02300389
Title: Randomized, Multi-center Clinical Trial Comparing Hypofractionated Radiotherapy Boost to Conventionally Fractionated in a High Risk Group of Prostate Cancer Patients
Brief Title: Comparing Hypofractionated Radiotherapy Boost to Conventionally Fractionated
Acronym: HYPOPROST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Greater Poland Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HYPOPROST
Record Dates: First submitted 2014-11-14; First posted 2014-11-25 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: high risk prostate cancer radiotherapy hypofractionation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated IMRT boost radiotherapy (Experimental): All patients included into this arm are irradiated to 46 Gy a 2 Gy fraction to the whole pelvis and seminal vesicles and prostate gland (I phase) and than the boost dose is limited to the prostate gland with some part of seminal vesicles with hypofractionated dose of 7.5 Gy in two fractions (II phase) to the total dose of 61 Gy. Additionally all patients received neoadjuvant Androgen Deprivation Therapy (3-4 months prior starting radiotherapy) and during radiotherapy and during the follow-up up to 24 months.
  Interventions: Radiation: Hypofractionated IMRT boost radiotherapy
- Conventional Fractionated IMRT boost radiotherapy (Active Comparator): All patients included into this arm are irradiated to 46 Gy a 2 Gy fraction to the whole pelvis and seminal vesicles and prostate gland (I phase) and than the boost dose is limited to the prostate gland with some part of seminal vesicles with conventional fractionated dose of 2 Gy in 15 fractions (II phase) to the total dose of 76 Gy. Additionally all patients received neoadjuvant Androgen Deprivation Therapy (3-4 months prior starting radiotherapy) and during radiotherapy and during the follow-up up to 24 months.
  Interventions: Radiation: Conventional Fractionated IMRT boost radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated IMRT boost radiotherapy — All patients included into this arm are irradiated to 46 Gy a 2 Gy fraction to the whole pelvis and seminal vesicles and prostate gland (I phase) and than the boost dose is limited to the prostate gland with some part of seminal vesicles with hypofractionated dose of 7.5 Gy in two fractions (II phase) to the total dose of 61 Gy. Additionally all patients received neoadjuvant Androgen Deprivation Therapy (3-4 months prior starting radiotherapy) and during radiotherapy and during the follow-up up to 24 months.
  Arms: Hypofractionated IMRT boost radiotherapy
Radiation: Conventional Fractionated IMRT boost radiotherapy — All patients included into this arm are irradiated to 46 Gy a 2 Gy fraction to the whole pelvis and seminal vesicles and prostate gland (I phase) and than the boost dose is limited to the prostate gland with some part of seminal vesicles with conventional fractionated dose of 2 Gy in 15 fractions (II phase) to the total dose of 76 Gy. Additionally all patients received neoadjuvant Androgen Deprivation Therapy (3-4 months prior starting radiotherapy) and during radiotherapy and during the follow-up up to 24 months.
  Arms: Conventional Fractionated IMRT boost radiotherapy

SUMMARY:
The main purpose of study is to compare the effectiveness of Hypofractionated IMRT boost Radiotherapy to Conventional IMRT boost Radiotherapy for high-risk prostate cancer patients combined with Androgen Deprivation Therapy.

DETAILED DESCRIPTION:
Additional objectives of the study for high-risk (non-metastatic) prostate cancer patients are as follows:

1. Analysis of number of circulating tumor cells in peripheral blood as a prognostic/predictive factors for survival.
2. Analysis of miRNA expression levels (100, 141 and 143) in peripheral blood as a prognostic and predictive factors.
3. Evaluation of the usefulness expression of selected proteins (PTEN, SMAD4, Cyclin D1, SPP1) as prognostic and predictive factors.
4. Evaluation of the usefulness of the expression level of antigen-specific T cells, B-and NK cells as a prognostic factors.
5. Evaluation of usefulness of the fiducial markers for localizing the prostate gland position during irradiation for the selected control imaging methods (2DkV, CBCT, MVCT).

ELIGIBILITY:
Inclusion Criteria:

* men from 40 to 75 years old with confirmed prostate adenocarcinoma, prostate biopsy will be performed <180 days before the date of randomization,
* completed assessment of tumor differentiation according to Gleason grading allows to perform stratification; Gleason score ≤ 7 versus Gleason score> 8,
* general condition according to the classification of the Eastern Cooperative Oncology Group (ECOG) 0 - 1), (Appendix 1),
* Androgen Deprivation Therapy: prior Radiotherapy (RT) (minimum 3 months before the start of RT), concurrently with RT and after RT during follow-up (24 months) ,
* high risk of Prostate Cancer progression defined as presence of at least one of the following factors: cT3, Gleason> 7, PSA> 20 ng / ml or presence of at least two of cT2c, Gleason 7, PSA in the range of 10.1 ng / ml to 19.9 ng / ml, cT defined by AJCC staging 7 edition, (Appendix 2),
* PSA identified at least 10 days after the biopsy or before, and patients receiving fiansteryd 30 days after the cessation of therapy,
* no regional and distant metastases confirmed by bone scintigraphy, chest radiograph, computed tomography/magnetic resonance imaging of the pelvis,
* signing an informed consent to participate in a medical experiment (radiotherapy + biological material samples) (Annex 3),
* morphological and biochemical parameters within normal limits.

Exclusion Criteria:

* the presence of active cancer except skin cancer preceding period of 5 years prior to randomization,
* Early surgery (radical prostatectomy) or pelvic RT,
* earlier hormonal therapy than is advocated in this study,
* co-morbidities that may significantly affect the expectancy life of the patients
* do not meet the criteria for inclusion.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2011-12; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
biochemical Progression Free Survival (bPFS) | 5 years
  Phoenix definition of biochemical failure

SECONDARY OUTCOMES:
Cause Specific Survival (CSS) | 5 years
  the period of time from randomization until death from prostate cancer
Overall Survival (OS) | 5years
  the period of time from randomization until death from any causes

OTHER OUTCOMES:
Toxicity of treatment | 5 years
  for toxicity of treatment RTOG classification is applied
Quality of Life (QOL) | 5 years
  for Quality of Life (QOL) the EORTC C30 and module PR25 is used.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Milecki, PhD., MD, Principal Investigator — Greater Poland Cancer Centre
Locations (3):
- Poland (3):
  - Lower-Silesian Oncology Centre, Wroclaw, Lower Silesian Voivodeship
  - Independent Public Healthcare of Ministry of Interior with Warmia and Mazury Oncology Centre, Olsztyn, Warmian-Masurian Voivodeship
  - Greater Poland Cancer Centre, Poznan, Wielkopolska

IPD SHARING:
Plan to Share IPD: No